CLINICAL TRIAL: NCT01236599
Title: Comparison of Polyethylene Wrap With and Without Previous Drying in Preterm Infants: A Randomized Clinical Trial.
Brief Title: Thermoregulation in the Preterm Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Luz María Cardona Torres, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LMCT-01
Record Dates: First submitted 2010-11-05; First posted 2010-11-08 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Nursing Care
Keywords: preterm infant, thermoregulation, polyethylene bag
MeSH Terms: conditions — Premature Birth | interventions — Polyethylene; Body Temperature Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- traditional care (No Intervention): Preterm Infants were placed under a radiant warmer (BLOSSON, Series 900, it Marks Fisher and Paykel), dried off and wrapped up in a sterile preheated field
  Interventions: Other: Polyethylene for thermoregulation in the preterm infant
- Polyethylene bag with previous drying (Experimental): infants were placed under the radiant warmer (BLOSSON, Series 900, it Marks Fisher and Paykel), dried off, and wrapped up in a polyethylene bag, leaving their faces discovered as well as the access at umbilical catheters or veined access.
  Interventions: Other: Polyethylene for thermoregulation in the preterm infant
- Polyethylene bag without previous drying (Experimental): Preterm infants were placed under a radiant warmer (BLOSSON, Series 900, it Marks Fisher and Paykel) and without previous body drying (only the head was dried), were wrapped up with the polyethylene bag, leaving their faces discovered as well as the access to umbilical catheters or veined access
  Interventions: Other: Polyethylene for thermoregulation in the preterm infant

INTERVENTIONS:
Other: Polyethylene for thermoregulation in the preterm infant — 3 groups with 30 preterm infants (PI) each one: 1) PI under radiant warmer, drying, wrapped in sterile field preheated (traditional care), 2) PI under radiant warmer, wrapped in polyethylene bag after drying, with their naked face and access to umbilical catheters or venous access, and 3) PI under radiant warmer, without drying, wrapped in polyethylene bag, with their naked face and access to umbilical catheters or venous access. Body temperature (BT) and incubator temperature (IT) were measured every 15 minutes from birth until 120 minutes of extra uterine life.
  Other Names: Heart loss in the preterm infant

SUMMARY:
The purpose of this study is to compare the response of temperature adaptation in preterm infant using the polyethylene wrap with and without previous drying.

DETAILED DESCRIPTION:
Preterm infants (PI) are predisposed to loss heat and have little subcutaneous tissue and a high ratio between surface and body weight and a reduced amount of glycogen deposits and brown fat (Gomella, 2005, p. 43).

In Mexico and South America in 2003 were reported 207.753 neonatal deaths, 21.4 per every 1,000 born alive in whom hypothermia was significant among infants with low birth weight and preterm infants. (Zuleta, Gomez & Jaramillo, 2009).

PRETERM INFANT Official Mexican Norm -007-SSA2-1993 (1995) considers a preterm infant as the product of the conception from 28-37 weeks of gestation, and weighing 1000-2499 g.

THERMOREGULATION OF PRETERM INFANT Survival of the newborn increases if the excessive loss heat is prevented. To achieve this purpose the newborn should be kept in a thermal environment neutral "which is what allows an infant consume the least amount of energy to maintain normal body temperature". (Karlsen, 2006, p. 49) The heat is gained or lost by convection 37% (between a child and a fluid: air stream or during bathing), conduction 4% (between two bodies in contact with different temperatures: the fields, mattress) radiation, 43% (between two solid surfaces that are not in touch: cool walls of the incubator) and 16% evaporation (heat loss in the conversion of water from liquid to gas, skin, breathing, sweating). (Tamez & Pantoja, 2004, pp. 29-30; Ruíz, 2007) The understanding of these forms of heat exchange provides the scientific basis for nursing interventions aimed at modifying the environment.

Response to cold stress of preterm infant: When the sensors of central and peripheral temperature detect stress for cold, they send signals to the hypothalamus. The hypothalamus activates the liberation of norepinephrine. This hormone causes increment in the metabolism, which increases the oxygen consumption and glucose utilization. The increment in the consumption of oxygen can induce hypoxemia and if it is severe, could progress to hypoxia. Peripheral vasoconstriction is limited in infant of very low birth weight in the first 48 hours of life; this increases the heat loss to level of the skin. In the preterm infant the loss heat occurs faster than its ability to produce and conserve heat. (Karlsen, 2006, p. 56) Adverse effects of cold stress in term and preterm neonate: When a term or a preterm neonate is hypothermic, the metabolism, oxygen consumption and glucose utilization increase. If the neonate, is experiencing trouble for breath, he will not be able of confront the increment in the demand of oxygen for tissues. This allows or increases the hypoxemia, which contributes to increased pulmonary vasoconstriction. The severe hypoxemia can progress to hypoxia, which leads to anaerobic metabolism. During anaerobic metabolism, the accumulation of lactic acid and blood ph drops is observed. If it is not reversed, the risk of death is high. (Jasso, 2005, p. 91; Karlsen, 2006, p. 58) The hypothermia can cause hypoglycemia, since the glucose is the primary source energy for the brain. The level of conscience of the neonate can diminish, the respiration can become slow and oxygenation will be affected. The survivors to an event of hypothermia have collateral effects as the increase of the difficulty of respiration, severe renal failure, disseminated coagulation, increase in the incidence of infection and persistence of the arterial conduit. (Karlsen, 2006, p. 58) PLACEMENT OF POLYETHYLENE BAG The program STABLE (sugar, temperature, airway, blood pressure, lab work and emotional support) for care post-resuscitation and pre-transport of sick neonates, recommended cover to premature infant with a plastic cover immediately after birth, from the neck down to reduce heat loss through evaporation and convection. (Karlsen, 2006, pp. 51, 53) The polyethylene bag, "is a cheap device, practical, simple, does not interfere with the immediate care or resuscitation (Vohra et al., 2004) and does not put in risk the integrity and security of the newborn. But it is not clear whether its effectiveness is similar with or without prior drying of the newborn, because the only study comparing these two techniques was conducted in term infants and it was not randomized (Menesses et al., 2002).

It is recommended that all apnea at birth should be treated as a secondary apnea and not delays resuscitation. (American Academy of Pediatrics and American Heart Association, 2000) At this stage every second is vital for the newborn, and from this comes the concern of knowing if the polyethylene bag is equally effective for thermoregulation of the newborn, with or without pre-drying, since it would save a few seconds for drying, and immediately beginning neonatal resuscitation.

ELIGIBILITY:
Inclusion Criteria:

Preterm Infant were included according with the Official Mexican Norm -007-SSA2-1993 (1995)

Exclusion Criteria:

* Preterm Infant were not included in case of malformations that involved lost of the cutaneous integrity or in case of severe cardiac congenital disease.

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Corporal temperature of preterm infants and Temperature of the incubator. | every 15 minutes until the two hours of extrauterine life
  Corporal temperature. An axillary thermometer of mercury was used, which was placed in the boy's armpit, making sure that it was in contact with the skin, during five minutes.
  Temperature of the incubator. It was directly registered from the incubator thermometer (medix TR 306). All the incubators started with a temperature of 34oC, and they were adjusted according to the necessity of preterm infant, when valuing the axillary temperature.

SECONDARY OUTCOMES:
Gestational age | . It was valued at birth by Capurro's score
  , the children from 28 to 37 weeks of gestational age that fulfilled the other inclusion approaches continued in the study. The Capurro's score considers five somatic data: nipple formation, skin texture, ear forms, breast nodule and plantar skin creases. First a partial punctuation was obtained considering each parameter, then the following formula was applied: (204 + partial punctuation) / 7 = gestational age
Weight | It was valued at birth
  . It was measured at birth with the PI naked using mechanical weighing machine
Apgar score | the minute and the five minutes of life
  Each one of the five identifiable characteristics with easiness was valued: muscle tone, heart rate, reflex irritability, skin coloration, breathing rate and effort, and each factor was scored on a scale of zero to two, the total punctuation, was determined with base in the sum of the five components
Heart rate | It was valued at birth and every 15 minutes until the two hours of extrauterine life
  using a stethoscope with a neonatal bell (Riester model luxe duplexR Marks) during 15 seconds, the result was multiplied for four, to obtain the heart frequency in one minute.
Breathing frequency | . It was valued at birth and every 15 minutes until the two hours of extrauterine life.
  The thoracic movements were observed during 30 seconds, considering the complete breathing cycle (inspiration and expiration). The obtained result was multiplied for two, to obtain the breathing frequency in one minute.
Capillar glucose | . It was measured at birth and at two hours of extrauterine life
  with the Optium Xceed monitor using ribbons of glucose test in blood (MediSense Optium).
Environmental temperature | It was registered at birth
  in the delivery room with an environmental thermometer (RadioShackR)
Blood pressure | . It was measured at 15 minutes, one hour and two hours of extrauterine life
  . It was valued by the flushing technique with a sphygmomanometer (Riester marks). The sphygmomanometer cuff was applied to the wrist or ankle and the distal portion of the extremity was compressed by firmly wrapping a wide, soft rubber drain around it, beginning at the tips of the digits and working proximally to the cuff edge. The manometer was rapidly inflated to 80 mmHg and the elastic wrapping removed. With gradual release of the pressure, a point was reached at which there was a distinct blush of the blanched portion of the extremity.

CONTACTS AND LOCATIONS:
Overall Officials: Norma Amador, PhD, Study Director — Instituto Mexicano del Seguro Social
Locations (1):
- Hospital General de Zona N 4. Instituto Mexicano del Seguro Social, Celaya, Guanajuato, Mexico

REFERENCES:
- [Background] Duman N, Utkutan S, Kumral A, Koroglu TF, Ozkan H. Polyethylene skin wrapping accelerates recovery from hypothermia in very low-birthweight infants. Pediatr Int. 2006 Feb;48(1):29-32. doi: 10.1111/j.1442-200X.2006.02155.x. PMID 16490066
- [Background] Lenclen R, Mazraani M, Jugie M, Couderc S, Hoenn E, Carbajal R, Blanc P, Paupe A. [Use of a polyethylene bag: a way to improve the thermal environment of the premature newborn at the delivery room]. Arch Pediatr. 2002 Mar;9(3):238-44. doi: 10.1016/s0929-693x(01)00759-x. French. PMID 11938534
- [Background] Vohra S, Roberts RS, Zhang B, Janes M, Schmidt B. Heat Loss Prevention (HeLP) in the delivery room: A randomized controlled trial of polyethylene occlusive skin wrapping in very preterm infants. J Pediatr. 2004 Dec;145(6):750-3. doi: 10.1016/j.jpeds.2004.07.036. PMID 15580195